CLINICAL TRIAL: NCT00550992
Title: International Collaborative Treatment Protocol for Infants Under One Year With Acute Lymphoblastic or Biphenotypic Leukemia
Brief Title: Different Therapies in Treating Infants With Newly Diagnosed Acute Leukemia
Acronym: Interfant06
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dutch Childhood Oncology Group (Other)
Collaborators: BFM Germany (Unknown); CORS Monza Italy (Unknown); Associazione Italiana Ematologia Oncologia Pediatrica (Other); Australian and New Zealand Children's Oncology Group (Other); BFM Austria (Unknown); CLCG France Belgium Portugal (Unknown); COALL Germany (Unknown); CPH, Czech republic (Unknown); DFCI consortium USA (Unknown); FRALLE France (Unknown); Hong Kong Government (Other Government); MD Anderson USA (Unknown); NOPHO Scandinavian countries (Unknown); PINDA, Chile (Unknown); PPLLSG Poland (Unknown); Seattle USA (Unknown); SJCRH USA (Unknown); UKCCSG United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000570260; DCOG-INTERFANT-06; EUDRACT-2005-004599-19; CCLG-LK-2006-10
Record Dates: First submitted 2007-10-22; First posted 2007-10-30 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; acute undifferentiated leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Biphenotypic, Acute | interventions — Antilymphocyte Serum; Asparaginase; Busulfan; Cyclophosphamide; Cyclosporine; Cytarabine; Daunorubicin; Etoposide; Leucovorin; Melphalan; Mercaptopurine; Methotrexate; Mitoxantrone; pegaspargase; Prednisolone; Prednisone; Hydrocortisone; Thioguanine; Vincristine; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: asparaginase
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: leucovorin calcium
Drug: melphalan
Drug: mercaptopurine
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: pegaspargase
Drug: prednisolone
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: thioguanine
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine, methotrexate, leucovorin, and antithymocyte globulin before and after transplant may stop this from happening. It is not yet known which treatment regimen is most effective in treating acute leukemia.

PURPOSE: This randomized clinical trial is studying how well different therapies work in treating infants with newly diagnosed acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare an early intensification regimen comprising two "acute myeloid leukemia" induction therapy blocks with a standard protocol IB regimen administered directly after induction therapy in medium-risk (MR) and high-risk (HR) patients with newly diagnosed acute lymphoblastic or biphenotypic leukemia.

Secondary

* To compare through a randomized study the role of these regimens in treating these patients.
* To compare the overall outcome of the Interfant-06 study with outcomes in the historical control series, especially in the Interfant-99 study.
* To compare the outcomes of low-risk, MR, or HR patients in this study with those of patients in the historical control series Interfant-99 study.
* To study which factors have independent prognostic value in patients treated with these regimens.
* To assess the role of stem cell transplantation in HR patients.

OUTLINE: This is a multicenter study.

* Induction therapy:

  * Prednisone phase: Patients receive prednisone orally or IV three times daily on days 1-7 and methotrexate (MTX) and prednisolone (PRDL) intrathecally (IT) on day 1. Patients then proceed to remission induction therapy.
  * Remission induction phase: Patients receive dexamethasone (DEXA) IV or orally three times daily on days 8-28 followed by a taper to 0 over 1 week; vincristine (VCR) IV on days 8, 15, 22, and 29; cytarabine (ARA-C) IV over 30 minutes on days 8-21; daunorubicin hydrochloride (DNR) IV over 1 hour on days 8 and 9; asparaginase (ASP) IV over 1 hour or intramuscularly (IM) on days 15, 18, 22, 25, 29, and 33; MTX IT on days 1 and 29*; and ARA-C IT on day 15. Patients also receive PRDL or therapeutic hydrocortisone (HC) IT on days 1, 15, and 29.

NOTE: *Patients with CNS involvement at initial diagnosis also receive MTX IT on days 8 and 22. If CNS leukemia is still present at day 29, then patients receive weekly MTX IT until the CNS is free of leukemia.

After completion of induction therapy, patients are stratified according to risk group (low-risk [LR] vs medium-risk [MR] vs high-risk [HR]). Patients with low-risk disease are assigned to treatment arm I. Patients with MR or HR disease that is in complete remission (CR) on day 33 are randomized to 1 of 2 treatment arms. These patients are stratified according to status (MR with rearranged MLL vs MR with unknown MLL vs HR).

* Arm I (standard therapy):

  * Protocol IB therapy (beginning on day 36 of induction therapy): Patients receive cyclophosphamide (CPM) IV over 1 hour on days 1 and 29 and oral mercaptopurine (MP) on days 1-28; ARA-C IV on days 3-6, 10-13, 17-20, and 24-27; ARA-C IT on day 10; and MTX IT on day 24. Patients also receive PRDL or therapeutic HC IT on days 10 and 24.
  * MARMA therapy:

    * Part I: Patients receive oral MP once daily on days 1-14; high-dose (HD) MTX IV over 24 hours on days 1 and 8; leucovorin calcium orally or IV at 42, 48, and 54 hours after each dose of MTX until MTX plasma levels are safe; and MTX IT on days 2 and 9. Patients also receive PRDL or therapeutic HC IT on days 2 and 9.
    * Part II: Patients receive HD ARA-C IV over 3 hours twice daily with 12-hour intervals on days 15, 16, 22, and 23; and pegaspargase (PEG-ASP) IV over 1 hour or IM on day 23.
  * OCTADA(D) reinduction therapy:

    * Part I: At least 2 weeks after the completion of MARMA chemotherapy, patients receive oral dexamethasone (DEXA) three times daily on days 1-14, followed by a taper to 0 at day 21; oral thioguanine (TG) once daily on days 1-28; VCR IV on days 1, 8, 15, and 22; DNR IV over 1 hour on days 1, 8, 15, and 22; PEG-ASP IV over 1 hour or IM on day 1; ARA-C IV on days 2-5, 9-12, 16-19, and 23-26; and ARA-C IT on days 1 and 15. Patients also receive PRDL or therapeutic HC IT on days 1 and 15.
    * Part II: Patients receive oral TG once daily on days 36-49; ARA-C IV once daily on days 37-40 and 45-48; and CPM IV over 1 hour on days 36 and 49.
  * Maintenance therapy: At least 2 weeks after completion of the last course of OCTADA(D) chemotherapy, patients receive oral MP once daily; oral MTX once weekly; MTX IT in weeks 1 and 15; and ARA-C IT in week 8. Patients also receive PRDL or therapeutic HC IT in weeks 1, 8, and 15. Treatment continues for up to 104 weeks after initial diagnosis in the absence of disease progression or unacceptable toxicity.
* Arm II (experimental therapy):

  * ADE therapy (beginning on day 36 of induction therapy: Patients receive ARA-C IV every 12 hours on days 1-10; DNR IV over 1 hour on days 1, 3, and 5; etoposide (VP-16) IV over 4 hours on days 1-5; and ARA-C IT on day 1. Patients also receive PRDL or therapeutic HC IT on day 1.
  * MAE therapy: Patients receive ARA-C IV every 12 hours on days 1-10; mitoxantrone hydrochloride IV over 1 hour on days 1, 3, and 5; VP-16 IV over 4 hours on days 1-5; and MTX IT on day 1. Patients also receive PRDL or therapeutic HC IT on day 1.
  * MARMA therapy:

    * Part I: Patients receive oral MP once daily on days 1-14; high-dose (HD) MTX IV over 24 hours on days 1 and 8; leucovorin calcium orally or IV at 42, 48, and 54 hours after each dose of MTX until MTX plasma levels are safe; and MTX IT on days 2 and 9. Patients also receive PRDL or therapeutic HC IT on days 2 and 9.
    * Part II: Patients receive HD ARA-C IV over 3 hours twice daily with 12-hour intervals on days 15, 16, 22, and 23; and pegaspargase (PEG-ASP) IV over 1 hour or IM on day 23.
  * OCTADA reinduction therapy:

    * Part I: At least 2 weeks after the completion of MARMA chemotherapy, patients receive oral DEXA three times daily on days 1-14, followed by a taper to 0 at day 21; oral TG once daily on days 1-28; VCR IV on days 1, 8, 15, and 22; PEG-ASP IV over 1 hour or IM on day 1; ARA-C IV on days 2-5, 9-12, 16-19, and 23-26; and ARA-C IT on days 1 and 15. Patients also receive PRDL or therapeutic HC IT on days 1 and 15.
    * Part II: Beginning 1 week after completion of part I, patients receive oral TG once daily on days 36-49; ARA-C IV once daily on days 37-40 and 45-48; and CPM IV over 1 hour on days 36 and 49.
  * Maintenance therapy: At least 2 weeks after completion of the last course of OCTADA chemotherapy, patients receive oral MP once daily; oral MTX once weekly; MTX IT in weeks 1 and 15; and ARA-C IT in week 8. Patients also receive PRDL or therapeutic HC IT in weeks 1, 8, and 15. Treatment continues for up to 104 weeks after initial diagnosis in the absence of disease progression or unacceptable toxicity.

All HR patients with a suitably matched donor are scheduled for allogeneic stem cell transplantation (SCT) after MARMA or before or during OCTADA(D) chemotherapy, provided they are in CR1 and no more than 8 months have elapsed since initial diagnosis.

* Conditioning regimens for allogeneic SCT:

  * Matched sibling donor (MSD): Patients receive oral busulfan (BU) every 6 hours on days -7 to -4; CPM IV over 1 hour on days -3 to -2; and melphalan (MEL) IV over 1 hour on day -1.
  * Matched donors (MD): Patients receive oral BU every 6 hours on days -7 to -4; CPM IV over 1 hour on days -3 to -2; MEL IV over 1 hour on day -1; and anti-thymocyte globulin (ATG) IV over 4 hours on days -3 to -1.
* Graft-Versus-Host Disease (GVHD) prophylaxis and therapy:

  * MSD: Patients receive cyclosporine (CsA) IV or orally twice daily beginning on day -1 and continuing to day 60 after SCT, followed by a taper in the absence of GVHD symptoms.
  * MD: Patients receive CsA as in group MSD; MTX IV on days 1, 3, and 6; leucovorin calcium IV on days 2, 4, and 7; and ATG IV on days -3 to -1.
* Allogeneic SCT: Patients undergo infusion of bone marrow, peripheral blood, or cord blood hematopoietic stem cells on day 0.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL) or biphenotypic leukemia meeting the following criteria:

  * Based on European Group for the Classification of Acute Leukemia (EGIL) diagnostic criteria
  * Newly diagnosed disease
  * Verified by morphology and confirmed by cytochemistry and immunophenotyping

    * Trephine biopsy is recommended (unless diagnosis can be confirmed by peripheral blood examination) in the event that bone marrow aspiration results in a "dry tap"
* Must have MLL gene rearrangements documented by split-signal fluorescence in situ hybridization and meets 1 of the following risk criteria:

  * Low-risk disease, defined as all MLL germline cases
  * Medium-risk disease, defined by 1 of the following criteria:

    * MLL status unknown
    * MLL rearranged AND age > 6 months
    * MLL rearranged AND age < 6 months AND WBC < 300 x 10^9/L AND prednisone good response
  * High-risk disease, defined by MLL rearrangement AND meets the following criteria:

    * Age at diagnosis < 6 months (i.e., < 183 days)
    * WBC ≥ 300 x 10^9/L AND/OR prednisone poor response
* Minimum donor and stem cell requirements for high-risk patients undergoing stem cell transplantation:

  * Donor meeting 1 of the following criteria:

    * HLA-identical sibling
    * Very well-matched related or unrelated donor
    * Must be HLA compatible in 10/10 or 9/10 alleles by 4 digit/allele high-resolution molecular genotyping
  * Stem cell source

    * Bone marrow (preferred source) OR peripheral blood stem cells of filgrastim [G-CSF]-stimulated donors OR cord blood

      * Highly-matched unrelated umbilical cord blood (UCB) (> 7/8 matches identified by high-resolution typing) accepted if a sibling donor is not able to donate bone marrow AND UCB with a sufficient number of nucleated cells (NCs) (i.e., > 1.5 x 10^7/kg recipient body weight [BW]) is cryopreserved
  * Must have ≥ 3 x 10^8 NCs/kg BW OR 3 x 10^6/kg BW CD34-positive cells available for transplantation
* CNS or testicular leukemia at diagnosis allowed

Exclusion criteria:

* Mature B-ALL, defined by the immunophenotypical presence of surface immunoglobulins or t(8;14) and breakpoint as in B-ALL
* Presence of the t(9;22) (q34;q11) or bcr-abl fusion in the leukemic cells (if data are not known, patient still may be eligible)
* Relapsed ALL

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior systemic corticosteroids

  * Corticosteroids by aerosol are allowed

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 445 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Survival
Event-free survival
Event-free survival within each risk group (i.e., low-risk, medium-risk, or high-risk)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Pieters, MD, MSC, PhD, Study Chair — Prinses Maxima Centrum voor kinderoncologie Utrecht; Martin Schrappe, MD, PhD, Study Chair — University Hospital Schleswig-Holstein
Locations (13):
- United States (4):
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- St. Anna Children's Hospital, Vienna, Austria
- Hopital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium
- University Hospital Motol, Prague, Czechia
- CHR Hotel Dieu, Nantes, France
- Germany (2):
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Nuovo Ospedale San Gerardo at University of Milano-Bicocca, Monza, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Great Ormond Street Hospital for Children, London, England, United Kingdom

REFERENCES:
- [Derived] Stutterheim J, van der Sluis IM, de Lorenzo P, Alten J, Ancliffe P, Attarbaschi A, Brethon B, Biondi A, Campbell M, Cazzaniga G, Escherich G, Ferster A, Kotecha RS, Lausen B, Li CK, Lo Nigro L, Locatelli F, Marschalek R, Meyer C, Schrappe M, Stary J, Vora A, Zuna J, van der Velden VHJ, Szczepanski T, Valsecchi MG, Pieters R. Clinical Implications of Minimal Residual Disease Detection in Infants With KMT2A-Rearranged Acute Lymphoblastic Leukemia Treated on the Interfant-06 Protocol. J Clin Oncol. 2021 Feb 20;39(6):652-662. doi: 10.1200/JCO.20.02333. Epub 2021 Jan 6. PMID 33405950
- [Derived] Pieters R, De Lorenzo P, Ancliffe P, Aversa LA, Brethon B, Biondi A, Campbell M, Escherich G, Ferster A, Gardner RA, Kotecha RS, Lausen B, Li CK, Locatelli F, Attarbaschi A, Peters C, Rubnitz JE, Silverman LB, Stary J, Szczepanski T, Vora A, Schrappe M, Valsecchi MG. Outcome of Infants Younger Than 1 Year With Acute Lymphoblastic Leukemia Treated With the Interfant-06 Protocol: Results From an International Phase III Randomized Study. J Clin Oncol. 2019 Sep 1;37(25):2246-2256. doi: 10.1200/JCO.19.00261. Epub 2019 Jul 8. PMID 31283407